CLINICAL TRIAL: NCT05071053
Title: Open-label Study of Tusamitamab Ravtansine (SAR408701) in Combination With Ramucirumab in Participants Previously Treated for Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma With CEACAM5-positive Tumors
Brief Title: Tusamitamab Ravtansine (SAR408701) in Combination With Ramucirumab in Pretreated Participants With Gastric Cancer
Acronym: CARMEN-GC01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, the decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT16444; U1111-1266-5040 (Registry Identifier: ICTRP); 2021-001967-26 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Adenocarcinoma Gastric; Gastrooesophageal Cancer
MeSH Terms: interventions — Ramucirumab; tusamitamab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tusamitamab ravtansine+Ramucirumab (Experimental): Participants received ramucirumab 8 milligram/kilogram (mg/kg) via intravenous (IV) infusion followed by tusamitamab ravtansine loading dose at 170 mg/meter square (m^2) via IV infusion on Cycle 1 Day 1 (each cycle was 2 weeks); and then ramucirumab 8 mg/kg via IV infusion followed by tusamitamab ravtansine 100 mg/m^2 via IV infusion at Cycle 2 and every 2 weeks (Q2W) in all subsequent cycles until disease progression, unacceptable adverse event (AE), death, initiation of a new anticancer therapy, or the participant's or investigator's decision to stop the treatment.
  Interventions: Drug: Ramucirumab (CYRAMZA®); Drug: Tusamitamab ravtansine (SAR408701)

INTERVENTIONS:
Drug: Ramucirumab (CYRAMZA®) — Pharmaceutical Form: Concentrate for solution for infusion
  Route of Administration: Intravenous Infusion
Drug: Tusamitamab ravtansine (SAR408701) — Pharmaceutical Form: Concentrate for solution for infusion
  Route of Administration: Intravenous Infusion

SUMMARY:
Primary Objectives:

Part 1: to confirm the recommended tusamitamab ravtansine loading dose Q2W in combination with ramucirumab in advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma population

Part 2: to assess the antitumor activity of tusamitamab ravtansine loading dose Q2W in combination with ramucirumab in advanced gastric or GEJ adenocarcinoma

Secondary Objectives:

* To assess safety and tolerability
* To assess durability of response (DOR)
* To assess progression-free survival (PFS)
* To assess the disease control rate (DCR)
* To assess the pharmacokinetics (PK)
* To assess the immunogenicity

DETAILED DESCRIPTION:
34 weeks (up to 4 weeks for screening, a median of 18 weeks for treatment, and a median of 12 weeks for end-of-treatment assessments and the safety follow-up visit).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of gastric or GEJ adenocarcinoma
* Metastatic disease or locally advanced, unresectable disease
* Participants who have measurable target lesion
* Participants with high carcinoembryonic antigen-related cell adhesion molecule (CEACAM5) expression as per central assessment on tumor biospsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Female participant who agrees to use effective contraceptive methods during and for at least 7 months after the last dose of treatment administration
* Male participant who agrees to use effective contraception methods during and for at least 4 months after the last dose of treatment administration
* Signed informed consent

Exclusion Criteria:

* Untreated brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression
* Significant concomitant illness
* History within the last 3 years of an invasive malignancy other than that treated in this study
* Known uncontrolled infection
* Nonresolution of any prior treatment-related toxicity
* Unresolved corneal disorder or any previous corneal disorder considered by an ophthalmologist to predict higher risk of drug-induced keratopathy
* Use of contact lenses
* Radiographic evidence of major airway or blood vessel invasion or intratumor cavitation
* History of uncontrolled hereditary or acquired thrombotic disorder or history of aneurism
* Major surgery within 28 days prior to Day 1/first IMP infusion; subcutaneous venous access device placement within 7 days prior to Day 1; or postoperative bleeding complications or wound complications from a surgical procedure performed in the last 2 months
* History of gross hemoptysis (defined as bright red blood or ≥1/2 teaspoon) within 2 months before the first treatment administration
* Any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months before the first administration of treatment administration
* Uncontrolled arterial hypertension (systolic ≥150 mmHg or diastolic ≥90 mmHg) despite standard medical management.
* Serious or nonhealing wound, skin ulcer, or bone fracture within 28 days before the first administration of treatment administration
* Gastrointestinal (GI) perforation and/or fistulae within 6 months prior to first administration of treatment administration
* Significant bleeding disorders, vasculitis, or Grade 3-4 gastrointestinal (GI) bleeding within 3 months before the first administration of study intervention.
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection Crohn's disease, ulcerative colitis, or chronic diarrhea
* Medical condition requiring concomitant administration of a medication with a narrow therapeutic window and metabolized by CYP450 or a strong CYP3A inhibitor
* Concurrent treatment with any other anticancer therapy
* Prior treatment targeting CEACAM5 or containing maytansinoid DM1 or DM4 or ramucirumab or taxane or targeting VEGF/VEGFR Poor organ function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- Belgium (3):
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560003, Edegem
  - Investigational Site Number : 0560001, Leuven
- Japan (4):
  - Investigational Site Number : 3920002, Kashiwa-shi, Chiba
  - Investigational Site Number : 3920004, Matsuyama, Ehime
  - Investigational Site Number : 3920001, Sapporo, Hokkaido
  - Investigational Site Number : 3920003, Sunto-gun, Shizuoka
- Russia (2):
  - Investigational Site Number : 6430003, Pushkin, Saint- Petersburg, Sankt-Peterburg
  - Investigational Site Number : 6430001, Arkhangelsk
- South Korea (4):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
- Spain (4):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Granada
  - Investigational Site Number : 7240001, Madrid
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920003, Ankara
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920004, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 investigational sites in 6 countries. A total of 45 participants were screened from 16-Nov-2021 to 17-Feb-2023 of which 10 were screen failures due to not meeting eligibility criteria. The study was terminated as per Sponsor decision and not related to any safety concern.
Pre-assignment Details: A total of 35 participants were enrolled in this study. All participants received the same dose in this single-group, single arm study as pre-specified in the protocol.
  Note: Reason for not completed = Reason for permanent full study intervention discontinuation.
Groups:
- Tusamitamab Ravtansine + Ramucirumab: Participants received ramucirumab 8 milligram/kilogram (mg/kg) via intravenous (IV) infusion followed by tusamitamab ravtansine loading dose at 170 mg/meter square (m^2) via IV infusion on Cycle 1 Day 1 (each cycle was 2 weeks); and then ramucirumab 8 mg/kg via IV infusion followed by tusamitamab ravtansine 100 mg/m^2 via IV infusion at Cycle 2 and every 2 weeks (Q2W) in all subsequent cycles until disease progression, unacceptable adverse event (AE), death, initiation of a new anticancer therapy, or the participant's or investigator's decision to stop the treatment.
Period: Overall Study
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Started (Enrolled) | 35
Completed (Treatment completion) | 0
Not Completed | 35
Not completed — Progressive disease | 30
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered.
Groups:
- Tusamitamab Ravtansine + Ramucirumab: Participants received ramucirumab 8 mg/kg via IV infusion followed by tusamitamab ravtansine loading dose at 170 mg/m^2 via IV infusion on Cycle 1 Day 1 (each cycle was 2 weeks); and then ramucirumab 8 mg/kg via IV infusion followed by tusamitamab ravtansine 100 mg/m^2 via IV infusion at Cycle 2 Q2W in all subsequent cycles until disease progression, unacceptable AE, death, initiation of a new anticancer therapy, or the participant's or investigator's decision to stop the treatment.
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Study-Drug Related Dose Limiting Toxicities (DLTs)
Description: The following AEs occurred during the first 2 cycles of treatment, unless due to disease progression or to a cause obviously unrelated to study drug, were considered DLTs:
  * Grade 4 neutropenia for 7 or more consecutive days.
  * Grade 3 to 4 neutropenia complicated by fever (temperature >=38.5 degree Celsius on more than 1 occasion) or microbiologically or radiographically documented infection.
  * Grade >=3 thrombocytopenia associated with clinically significant bleeding requiring clinical intervention.
  * Grade 4 non-hematologic AE.
  * Grade >=3 keratopathy. In addition, any other AE that the Investigators and sponsor deemed to be dose limiting, regardless of its grade, was also considered as DLT.
Time Frame: From Cycle 1 Day 1 to Cycle 2 Day 14; approximately 28 days
Population: DLT-evaluable population included all enrolled participants who received 2 cycles with at least 80% of the intended dose for both tusamitamab ravtansine and ramucirumab at each of the 2 first infusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as percentage of participants with confirmed complete response (CR) or partial response (PR) as best overall response (BOR) determined per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor assessments performed at Baseline (Day 1), then every 6 weeks (±7 days) thereafter, approximately 88.1 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 35
percentage of participants | 14.3 [4.81 to 30.26]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A SAE was defined as any untoward medical occurrence that, at any dose: resulted in death or was life-threatening or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent disability/incapacity or congenital anomaly/birth defect. TEAE was defined as AEs that developed, worsened, or became serious during the treatment-emergent period.
Time Frame: From the first study drug administration (Day 1) up to 30 days after the last study drug administration, approximately 120 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 35
Participants
  Any TEAE | 35
  Any TESAE | 15

4. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time from first documented evidence of CR or PR until progressive disease (PD) determined per RECIST v1.1 or death from any cause, whichever occured first. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Tumor assessments performed at Baseline (Day 1), then every 6 weeks (±7 days) thereafter, approximately 88.1 weeks
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. Only participants with confirmed CR or PR as BOR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 5
months | NA [5.520 to NA] — NA indicates that the median and upper limit of confidence interval (CI) were not estimable due to insufficient number of participants with events at study closure.

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The PFS was defined as the time from the first study drug administration to the date of the first documented disease progression or death due to any cause, whichever came first as per RECIST v1.1.
Time Frame: Tumor assessments performed at Baseline (Day 1), then every 6 weeks (±7 days) thereafter, approximately 88.1 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 35
months | 3.78 [1.511 to 5.749]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who achieved confirmed CR, confirmed PR or stable disease (SD) as per RECIST v1.1. The SD was defined as neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Tumor assessments performed at Baseline (Day 1), then every 6 weeks (±7 days) thereafter, approximately 88.1 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 35
percentage of participants | 62.9 [44.92 to 78.53]

7. Secondary Outcome: Individual Observed Predose Concentrations (Ctrough) of Tusamitamab Ravtansine
Description: Blood samples were collected for the measurement of Ctrough of tusamitamab ravtansine.
Time Frame: Pre-infusion on Cycle 2 Day 1
Population: The Pharmacokinetic (PK) population included all participants from the all-treated population with at least 1 post-baseline PK concentration (whatever the cycle and even if dosing was incomplete) with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at specified timepoint are reported.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 30
microgram/milliliter (mcg/mL) | 14.7 (6.83)

8. Secondary Outcome: Individual Observed Predose Concentrations (Ctrough) of Ramucirumab
Description: Blood samples were collected for the measurement of Ctrough of concentrations of ramucirumab.
Time Frame: Pre-infusion on Cycle 2 Day 1
Population: The PK population included all participants from the all-treated population with at least 1 post-baseline PK concentration (whatever the cycle and even if dosing was incomplete) with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at specified timepoint are reported.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 29
mcg/mL | 21.8 (10.48)

9. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATAs) Against Tusamitamab Ravtansine
Description: Blood samples were collected to assess the presence of ATA against tusamitamab ravtansine in plasma from all participants. ATA incidence was defined as the number of participants found to have seroconverted (treatment-induced ATAs) or boosted their pre-existing ATA response (treatment-boosted ATAs) at any time after first study drug administration.
Time Frame: Upto 92.1 weeks
Population: The ATA population included all participants from the all-treated population with at least 1 post-baseline ATA result (negative, positive, or inconclusive).
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
Number analyzed (Participants) | 31
Participants
  Treatment-induced ATA | 4
  Treatment-boosted ATA | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first study drug administration (Day 1) up to 30 days after the last study drug administration, approximately 120 weeks. All-cause mortality (death) was assessed from signing of the informed consent form to study termination, approximately 155 weeks.
Description: Analysis was performed on all-treated population. All participants received the same dose in this single-group, single arm study as pre-specified in the protocol.
Arm/Group | Tusamitamab Ravtansine + Ramucirumab
All-Cause Mortality (participants affected / at risk) | 13/35
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine + Ramucirumab (N=35)
Covid-19 (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Death (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine + Ramucirumab (N=35)
Covid-19 (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 5 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (11)
Decreased Appetite (Metabolism and nutrition disorders) | 8 (8)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (3)
Keratitis (Eye disorders) | 3 (4)
Keratopathy (Eye disorders) | 8 (13)
Vision Blurred (Eye disorders) | 3 (3)
Hypertension (Vascular disorders) | 10 (15)
Hypotension (Vascular disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 10 (12)
Nausea (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 3 (3)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 5 (9)
Asthenia (General disorders) | 5 (5)
Fatigue (General disorders) | 8 (9)
Oedema Peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (7)
Alanine Aminotransferase Increased (Investigations) | 4 (6)
Aspartate Aminotransferase Increased (Investigations) | 6 (8)
Neutrophil Count Decreased (Investigations) | 3 (8)
Platelet Count Decreased (Investigations) | 5 (9)

LIMITATIONS AND CAVEATS:
The study was terminated as per Sponsor decision and not related to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT05071053/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05071053/SAP_001.pdf